CLINICAL TRIAL: NCT04130347
Title: Acute Kidney Injury in Major Abdominal Surgery: Retrospective Study of 501 Patients
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Michael Hultström, Associate professor, Uppsala University
Other Study IDs: EPN dnr 2017/218
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Blood samples collected one year ahead of surgery and one year after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pancreatic resection
- Liver resection
- HIPEC surgery
- Gynecological debulking surgery

SUMMARY:
Retrospective study that aims to examine the presence of acute kidney injury (AKI) during major abdominal surgery, non- cardiac surgery. Using clinical and biochemical data in order to establish AKI frequency and risk factors.

DETAILED DESCRIPTION:
Ethical approval was submitted and approved by the regional ethical committee, Etisk prövningsnämnd Uppsala, # 2017/418.

Patients were selected from the time span of april 2016 to september 2017. The investigators identified 499 patients that had undergone any of the selected procedures. The procedures were, pancreatic resection, HIPEC surgery in colorectal setting, gynecological debulking in metastasized ovarian cancer, and liver resection.

The risk of acute kidney injury (AKI) by the KDIGO definition during the postoperative period will be estimated in the group as a whole, and for each type of surgery separately. In addition the data will be stratified by sex to investigate systematic gender disparities or physiological differences. Length of stay, thirty day and sixty day mortality will secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

Any of the selected procedures.

Exclusion Criteria:

Patient has expressed his or her will to nor participate in any study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Swedish population undergoing cancer surgery with four selected procedures. Age span between 19 and 85 years old.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI | the first 24- 72 hours postop
  Frequency of AKI as defined by KDIGO

SECONDARY OUTCOMES:
Mortality | 30, 60 and 360 days postoperatively
  30, 60, and 360 day mortality rate
Major Adverse Kidney Events | 30, 60 and 360 days postoperatively
  Renal composite outcome according to Major Adverse Kidney Events (MAKE)
Fluid balance | 24-72h
  Fluid balance during surgery, and the first postoperative days.
Electrolyte disturbances | 24-72h
  Any electrolyte disturbance.

IPD SHARING:
Plan to Share IPD: No